CLINICAL TRIAL: NCT01171352
Title: Predicting Hypotension During Dialysis in the ICU
Status: Withdrawn | Type: Observational
Why Stopped: Lack of funding
Sponsor: Oregon Health and Science University (Other)
Responsible Party: Sponsor
Other Study IDs: IRB00006189
Record Dates: First submitted 2010-07-27; First posted 2010-07-28 (Estimated); Last update posted 2019-06-05 (Actual); Status verified 2019-06

CONDITIONS: Peridialytic Hypotension
Keywords: hemodialysis; dialysis; hypotension; CritLine; PiCCO; Thermodilution; CVVHDF; IHD
MeSH Terms: conditions — Hypotension

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- ICU Dialysis Patients: Any patient 18 years and older who is admitted to the OHSU Hospitals ICUs with ARF, or End Stage Renal Disease (ESRD) for a diagnosis other than hyperkalemia, as the sole determinant for that level of care, will be invited to participate. The patient must have acute or chronic needs for dialytic support during their ICU stay.
  Interventions: Procedure: Transpulmonary Thermodilution

INTERVENTIONS:
Procedure: Transpulmonary Thermodilution — A PiCCO femoral catheter will be placed and PiCCO parameters will be obtained using transpulmonary thermodilution after continuous dialysis is ordered or just prior to initiation of intermittent dialysis, hourly until either completion of intermittent dialysis or 8 hours of continuous dialysis is completed.
  Other Names: Pulsion Medical Systems; PiCCO2; PiCCO

SUMMARY:
Currently, decisions regarding volume management for dialysis sessions in the ICU are made in large part on the nephrologists'/intensivists' overall gestalt. This gestalt is based upon a combination of commonly used measures of circulatory function, the physical exam, fluid balance, estimates of dialysis dry weight, and monitoring changes in relative blood volume status using devices such as the Crit-Line™ III, and central venous pressures. However, these tools perform poorly in predicting the circulatory system's overall response to dialysis. Consequently, episodes of dangerously low blood pressure are still frequently encountered. Better techniques to predict the circulatory system's response to dialysis are much needed. The intent of this study is to test newer metrics of circulatory system function for their ability to predict low blood pressure episodes during dialysis. This is important because it may enable the design of newer treatment strategies created to prevent low blood pressure episodes during dialysis and improve patient outcomes. The investigators overall hypothesis is that newer measures of vascular volume and dynamic indices of fluid responsiveness, previously found to better reflect cardiac preload state than currently used parameters, will better predict low blood pressure episodes during dialysis than current methods.

ELIGIBILITY:
Inclusion Criteria:

* Admitted to OHSU Hospitals ICUs
* Patient has acute or chronic needs for intermittent hemodialysis support during their ICU stay for any reason other than isolated hyperkalemia
* Central venous access in place separate from the dialysis catheter, or arteriovenous fistula or graft
* Two or more organ systems affected by critical illness requiring supportive care as documented in the medical chart.

Exclusion Criteria:

* age younger than 18 years old
* Weight > 160 kg
* burns greater than 40% total body surface area
* known cardiac or vascular aneurysm
* contraindications to femoral arterial puncture
* diagnosis of peripheral vascular disease
* not committed to full support
* participation in other experimental medication trial within 30 days
* current atrial or ventricular arrhythmias
* history of sever CHF- NYHA class >= III, previously documented EF < 30%
* severe aortic regurgitation
* anticipated ICU stay < 24 hrs
* not expected to require dialysis > 48 hours

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Any patient 18 years and older who is admitted to the OHSU Hospitals ICUs with ARF, or End Stage Renal Disease (ESRD) for a diagnosis other than hyperkalemia, as the sole determinant for that level of care, will be invited to participate. The patient must have acute or chronic needs for dialytic support during their ICU stay in order to qualify for the study. Dialysis support may be provided by intermittent HD sessions, or continuous venovenous hemodiafiltration (CVVHDF) depending on the underlying hemodynamic stability of the patient.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2010-07-19 (Actual); Primary Completion 2013-03-11 (Actual); Study Completion 2013-03-11 (Actual)

PRIMARY OUTCOMES:
hypotensive episode | during or within one hour post dialysis
  A mean arterial pressure of <60 mmHg, a 15% decrease from baseline systolic blood pressure at the start of the dialysis treatment regardless of modality, the need for fluid bolusing >7 mL/kg body weight, or initiation or increase of vasopressor medication in order to maintain MAP >60 mmHg.

SECONDARY OUTCOMES:
fluid removal tolerance | during the 4 hours following parameter measurement in dialysis
  Parameters measured will be examined to discriminate between patients that will tolerate fluid removal (UF) during the following 4 hours of dialysis if UF is ordered by physician (no hypotensive events with > 500 mL fluid removal) from those that won't
predicted volume of fluid that can be removed without hypotensive events | during dialysis
  Parameters measured will be examined to see if they can predict the volume of fluid successfully removed without hypotensive events
mortality in the ICU | duration of ICU stay
All cause mortality | 30 days
Length of stay in ICU | ICU stay duration
Length of stay in hospital | duration of hospital stay

CONTACTS AND LOCATIONS:
Overall Officials: Charles R Phillips, MD, Principal Investigator — Oregon Health and Science University
Locations (1):
- Oregon Health and Science University, Portland, Oregon, United States

REFERENCES:
- [Background] U.S. Renal Data System, USRDS 2008 Annual Data Report: Atlas of Chronic Kidney Disease and End-Stage Renal Disease in the United States. In: National Institutes of Health, National Institute of Diabetes and Digestive and Kidney Diseases, Bethesda, MD; 2008.
- [Background] Higgins TL, Teres D, Copes WS, Nathanson BH, Stark M, Kramer AA. Assessing contemporary intensive care unit outcome: an updated Mortality Probability Admission Model (MPM0-III). Crit Care Med. 2007 Mar;35(3):827-35. doi: 10.1097/01.CCM.0000257337.63529.9F. PMID 17255863
- [Background] Rocha E, Soares M, Valente C, Nogueira L, Bonomo H Jr, Godinho M, Ismael M, Valenca RV, Machado JE, Maccariello E. Outcomes of critically ill patients with acute kidney injury and end-stage renal disease requiring renal replacement therapy: a case-control study. Nephrol Dial Transplant. 2009 Jun;24(6):1925-30. doi: 10.1093/ndt/gfn750. Epub 2009 Jan 22. PMID 19164319
- [Background] Uchino S, Morimatsu H, Bellomo R, Silvester W, Cole L. End-stage renal failure patients requiring renal replacement therapy in the intensive care unit: incidence, clinical features, and outcome. Blood Purif. 2003;21(2):170-5. doi: 10.1159/000069156. PMID 12601260
- [Background] Daugirdas JT. Pathophysiology of dialysis hypotension: an update. Am J Kidney Dis. 2001 Oct;38(4 Suppl 4):S11-7. doi: 10.1053/ajkd.2001.28090. PMID 11602456
- [Background] Goedje O, Seebauer T, Peyerl M, Pfeiffer UJ, Reichart B. Hemodynamic monitoring by double-indicator dilution technique in patients after orthotopic heart transplantation. Chest. 2000 Sep;118(3):775-81. doi: 10.1378/chest.118.3.775. PMID 10988202
- [Background] Krepel HP, Nette RW, Akcahuseyin E, Weimar W, Zietse R. Variability of relative blood volume during haemodialysis. Nephrol Dial Transplant. 2000 May;15(5):673-9. doi: 10.1093/ndt/15.5.673. PMID 10809809
- [Background] Davenport A. Can advances in hemodialysis machine technology prevent intradialytic hypotension? Semin Dial. 2009 May-Jun;22(3):231-6. doi: 10.1111/j.1525-139X.2009.00614.x. PMID 19572996
- [Background] Sakka SG, Reinhart K, Meier-Hellmann A. Comparison of pulmonary artery and arterial thermodilution cardiac output in critically ill patients. Intensive Care Med. 1999 Aug;25(8):843-6. doi: 10.1007/s001340050962. PMID 10447543
- [Background] Michard F, Alaya S, Zarka V, Bahloul M, Richard C, Teboul JL. Global end-diastolic volume as an indicator of cardiac preload in patients with septic shock. Chest. 2003 Nov;124(5):1900-8. doi: 10.1378/chest.124.5.1900. PMID 14605066
- [Background] Michard F, Teboul JL. Predicting fluid responsiveness in ICU patients: a critical analysis of the evidence. Chest. 2002 Jun;121(6):2000-8. doi: 10.1378/chest.121.6.2000. PMID 12065368
- [Background] Phillips CR, Watters JM, Hagg DS, et al. Global end-diastolic volume as an indicator of cardiac preload in hemorrhagic shock and resuscitation in swine. Critical Care 2008;12(Suppl 2):P104.
- [Background] Phillips CR, Vinecore K, Hagg DS, Sawai RS, Differding JA, Watters JM, Schreiber MA. Resuscitation of haemorrhagic shock with normal saline vs. lactated Ringer's: effects on oxygenation, extravascular lung water and haemodynamics. Crit Care. 2009;13(2):R30. doi: 10.1186/cc7736. Epub 2009 Mar 4. PMID 19257901
- [Background] Michard F, Boussat S, Chemla D, Anguel N, Mercat A, Lecarpentier Y, Richard C, Pinsky MR, Teboul JL. Relation between respiratory changes in arterial pulse pressure and fluid responsiveness in septic patients with acute circulatory failure. Am J Respir Crit Care Med. 2000 Jul;162(1):134-8. doi: 10.1164/ajrccm.162.1.9903035. PMID 10903232
- [Background] De Backer D, Heenen S, Piagnerelli M, Koch M, Vincent JL. Pulse pressure variations to predict fluid responsiveness: influence of tidal volume. Intensive Care Med. 2005 Apr;31(4):517-23. doi: 10.1007/s00134-005-2586-4. Epub 2005 Mar 8. PMID 15754196
- [Background] Reddan DN, Szczech LA, Hasselblad V, Lowrie EG, Lindsay RM, Himmelfarb J, Toto RD, Stivelman J, Winchester JF, Zillman LA, Califf RM, Owen WF Jr. Intradialytic blood volume monitoring in ambulatory hemodialysis patients: a randomized trial. J Am Soc Nephrol. 2005 Jul;16(7):2162-9. doi: 10.1681/ASN.2004121053. Epub 2005 Jun 1. PMID 15930095